CLINICAL TRIAL: NCT01776411
Title: Phase I/II Clinical Study of Forodesine in Japanese Recurrent/Refractory Peripheral T-cell Lymphoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mundipharma K.K. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDS-J02
Record Dates: First submitted 2013-01-22; First posted 2013-01-28 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Recurrent or Refractory PTCL
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Experimental): Drug: forodesine hydrochloride 600 mg / body/day (3 x 100 mg capsules twice daily)
  Interventions: Drug: forodesine hydrochloride

INTERVENTIONS:
Drug: forodesine hydrochloride

SUMMARY:
Phase I portion:

To confirm safety and tolerability in recurrent/refractory peripheral T-cell lymphoma patients during repeated oral administration of forodesine 300 mg twice daily (600 mg/day) for 28 days, and determine the recommended dose. Also, to evaluate pharmacokinetics.

Phase II portion:

To evaluate the efficacy, safety, and pharmacokinetics of the recommended dosage regimen determined in the phase I portion. The primary efficacy endpoint shall be objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

* Japanese patients at least 20 years of age.
* Patients histologically diagnosed with peripheral T-cell lymphoma by pathological diagnosis of biopsied lesion. In this study, peripheral T-cell lymphoma is defined as the following mature T-cell/NK-cell neoplasms found in the 4th edition of the WHO Classification.
* Recurrent/refractory patients with a treatment history of at least one regimen.
* Patients with an enlarged lymph node or extranodal mass lesion clearly measurable in two perpendicular directions and greater than 1.5 cm in maximum diameter on computed tomography performed.
* Patients expected to survive for at least 3 months.
* ECOG PS 0-1.
* Patients with adequate hemopoietic efficacy, liver and kidney function.
* Patients from whom written consent has been obtained prior to study initiation.

Exclusion Criteria:

* Patients who received a chemotherapy agent or a high dose of a systemic adrenocorticosteroid within 21 days prior to initial administration of the study drug.
* Patients who received radiation therapy, phototherapy, or electron beam therapy within 21 days prior to initial administration of the study drug.
* Patients who received another study drug within 28 days prior to initial administration of the study drug.
* Patients who received antibody therapy within 100 days prior to initial administration of the study drug.
* Patients with a history of allogeneic hematopoietic stem cell transplantation. Or patients with a history of autologous hematopoietic stem cell transplantation within 100 days prior to initial administration of the study drug.
* Patients with cerebral metastasis or central nervous system lesion or a past history.
* Patients with active multiple primary cancer. Or patients with a history of a malignant neoplasm other than peripheral T-cell lymphoma within the past 5 years.
* Patients with severe cardiovascular disease.
* Patients with congenital long QT syndrome.
* Patients with QTcF >0.48 sec.
* Patients positive for HBs antigen, HCV antibody or HIV antibody on immunological investigation. Or patients positive for either HBc antibody or HBs antibody, and showing DNA more than sensitivity in HBV-DNA assay.
* Patients positive for CMV antigen on immunological investigation.
* Patients with infectious disease requiring treatment consisting of intravenous administration of antibacterial agent, fungicide, or antiviral drug.
* Patients with interstitial pneumonia or pulmonary fibrosis, or patients judged to have insufficient pulmonary function.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-03 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) based on evaluation by image assessment committee | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kensei Tobinai, MD,PhD, Principal Investigator — National Cancer Center Hospital
Locations (21):
- Japan (21):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Gunma University Hospital, Maebashi, Gunma
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - Tokai University Hospital, Isehara, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Osaka University Hospital, Suita, Osaka
  - Shimane University Hospital, Izumo, Shimane
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - National Cancer Center Hospital, Chūō, Tokyo
  - The Cancer Institute Hospital Japanese Foundation for Cancer Research, Koto, Tokyo
  - University of Fukui Hospital, Fukui
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Fukuoka University Hospital, Fukuoka
  - Imamura Bun-in Hospital, Kagoshima
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Okayama University Hospital, Okayama